CLINICAL TRIAL: NCT01490736
Title: Phase 1/2 Study of Photodynamic Therapy (PDT) With Lemuteporfin Topical Solution (LTS) in Healthy Volunteers and in Subjects With Mild Acne
Brief Title: Phase 1/2 Sequentially Staged Safety Study in Healthy Subjects and Subjects With Mild Acne
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dermira, Inc. (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: LTS ACN-05
Record Dates: First submitted 2011-12-07; First posted 2011-12-13 (Estimated); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Acne
Keywords: Acne; Sebum gland disease
MeSH Terms: conditions — Acne Vulgaris | interventions — lemuteporfin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- LTS/Vehicle (Experimental): Within subject control study
  Interventions: Drug: Lemuteporfin

INTERVENTIONS:
Drug: Lemuteporfin — lemuteporfin topical solution, 1%

SUMMARY:
The purpose of this study is to determine the safety of photodynamic therapy (PDT) with lemuteporfin topical solution (LTS) in healthy subjects and subjects with mild acne.

DETAILED DESCRIPTION:
This is a sequentially staged (Stage 1-4), proof of concept study assessing the safety of photodynamic therapy (PDT) and lemuteporfin topical solution (LTS) in healthy subjects and subjects with mild acne. Approximately 12 subjects will be enrolled in Stage 1 in order to determine a maximum tolerated light dose following LTS application. Up to 90 subjects with mild acne will be enrolled in Stage 2 in order to assess the safety of PDT following a single LTS application. Up to 50 subjects will be enrolled in Stage 3 in order to assess the safety of PDT following repeat LTS applications. Up to 40 subjects will be enrolled into Stage 4 to assess multiple treatments of LTS-PDT.

ELIGIBILITY:
Inclusion Criteria:

* Stage 1 only: healthy subjects
* Stage 1-4: male or female subjects age 18 years or older
* Stage 2: subjects with sebum excretion rate of 4 or higher on forehead
* Stage 2-4: subjects with at least 2 inflammatory acne lesions on the forehead
* Stage 3-4: subjects with sebum excretion rate of 5 or higher on forehead

Exclusion Criteria:

* Poor skin condition on back (Stage 1) or face (Stage 2 & 3)
* Severe facial acne, acne fluminans/conglobata, or nodulocystic acne
* Stage 2-4: previous use of Diane-35 within 6 months of Day 0, systemic acne treatment or systemic antibiotic treatment within 28 days of Day 0, topical acne treatment to the face within 14days of Day 0 or PDT to the face within 3 months of Day 0
* Stage 2-4: previous treatment of isotretinoin or other oral retinoids

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2011-12; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change in sebum excretion rate | Baseline to Day 14

SECONDARY OUTCOMES:
Change in biomarkers (e.g., caspase-3, CD163, neutrophil elastase) | Baseline to Day 14
Change in acne lesion count | Baseline to Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bissonnette, MD, Principal Investigator — Innovaderm Research Inc.
Locations (1):
- Innovaderm Research, Inc, Montreal, Quebec, Canada